

NCT05213390

30 August 2022

#### CENTRE FOR HEALTH TECHNOLOGY



EUR ING Edward Meinert MA MSc MBA MPA PhD CEng FBCS Associate Professor of eHealth

# Statistical analysis plan

## Using the variables:

- doraoutcomeupdate (0 = pass, no review, 1 = fail, needs review)
- supervisoroutcomeupdate (0 = pass, no review, 1 = fail, needs review)

# **Primary outcome:** Agreement between Dora and clinician for overall outcome decision and each symptom (x5)

- Inter-rater reliability (kappa)
- Accuracy (%)
- Data regarding true/false negatives/positives

| | Clinician: follow-up (1) | Clinician: no follow-up (0) |
|---|---|---|
| Dora: follow-up (1) | TP | FP |
| Dora: no follow-up (0) | FN | TN |

• Sensitivity, specificity, AUC

#### Secondary outcomes

# Clinical safety: Comparison with real complication rate

\*Note: please do this analysis three times, once for each of the three complication measures

• Data regarding true/false negatives/positives (**Tables 2-3**)

| | Complications: 3 month audit | No complications: 3 month audit |
|---|---|---|
| Dora: follow-up | ТР | FP |
| Dora: no follow-up | FN | TN |

- Sensitivity, specificity, AUC
- Variables
  - o Dora follow up: "doraoutcomeupdate"
  - Complications:
    - "hospital-review-within-3-months"
      - 0 = no hospital review, 1 = hospital review
    - "unexpected-change-management"
      - 0 = no unexpected change management, 1 = unexpected change management

# UNIVERSITY OF PLYMOUTH

## CENTRE FOR HEALTH TECHNOLOGY

EUR ING Edward Meinert MA MSc MBA MPA PhD CEng FBCS Associate Professor of eHealth

- "unplanned-hospital-rev"
  - 0 = no hospital review, 1 = hospital review